CLINICAL TRIAL: NCT01308892
Title: Cardiovascular Health Effects of Flavanol Rich Chocolate
Acronym: CHOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Wageningen universiteit department of human nutrition, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: NL33506.081.10
Record Dates: First submitted 2011-02-15; First posted 2011-03-04 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High flavaonol chocolate (Active Comparator)
  Interventions: Dietary Supplement: High flavanol chocolate; Dietary Supplement: High fat challenge
- Low flavanol chocolate (Placebo Comparator)
  Interventions: Dietary Supplement: Low flavanol chocolate; Dietary Supplement: High fat challenge

INTERVENTIONS:
Dietary Supplement: High flavanol chocolate — chocolate high in flavanols
  Arms: High flavaonol chocolate
Dietary Supplement: Low flavanol chocolate — chocolate low in flavanols
  Arms: Low flavanol chocolate
Dietary Supplement: High fat challenge — Milkshake with 95g fat

SUMMARY:
In the CHOC study the investigators will examine the effect of chocolate flavanols on vascular function, inflammation, oxidative stress and markers of endothelial function. The effects of both acute consumption and prolonged consumption will be studied. The secondary objectives are to investigate if daily intake of chocolate flavanols for 4 weeks will improve the response to a high fat/high energy challenge.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 45-70 years old
* BMI between 25 and 32 kg/m2

Exclusion Criteria:

* Urine glucose concentrations outside normal ranges (> 0,25 g/l)
* Fasting blood glucose < 7.0 mmol/L)
* Systolic Bp > 160 mmHg or diastolic Bp > 100 mmHg
* Blood Hb values below 8.4 mmol/L
* Allergic to cow milk, dairy products or chocolate
* Vegetarian
* Tobacco smoker
* Diagnosed with any long-term medical condition (e.g., diabetes, hemophilia, cardiovascular disease, anemia, gastrointestinal disease, renal failure)

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 0, 4wk
FMD | 0, 4wk
PWA | 0, 4wk

SECONDARY OUTCOMES:
leukocyte count and activation | 0, 4wk
PBMC gene expression | 0, 4wk
Markers of inflammation and ED | 0, 4wk
Blood pressure | 0 and 2h
  acute study part
FMD | 0 and 2hrs
  acute study part
PWA | 0 and 2 hrs
  acute study part
Leukocyte count and activation | 0 and 2 hrs
  acute study part
PBMC gene expression | 0 and 2 hrs
  acute study part
markers of inflammation and ED | 0 and 2hrs
  acute study part

CONTACTS AND LOCATIONS:
Overall Officials: Michael Müller, Prof.Dr, Study Chair — Chair Department of human nutrition NMG group
Locations (1):
- Wageningen universiteit division of human, Wageningen, Gelderland, Netherlands